CLINICAL TRIAL: NCT06937177
Title: Safely Optimizing Body Weight With TCMCB07 in Patients With Newly Diagnosed Metastatic Colorectal Cancer Undergoing Chemotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Endevica Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCMCB07-01
Record Dates: First submitted 2025-03-25; First posted 2025-04-22 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Cancer Weight Loss
Keywords: Metastatic colorectal cancer; Colorectal carcinoma; BMI; Weight Loss; Cachexia; Chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms; Weight Loss; Cachexia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study i.e. all study team members and study participants will remain blinded for the duration of the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo administered subcutaneously daily for 12 weeks (Placebo Comparator)
  Interventions: Drug: Placebo
- TCMCB07 12.5 mg administered subcutaneously daily for 12 weeks (Experimental)
  Interventions: Drug: TCMCB07
- TCMCB07 25 mg administered subcutaneously daily for 12 weeks (Experimental)
  Interventions: Drug: TCMCB07
- TCMCB07 50 mg administered subcutaneously daily for 12 weeks (Experimental)
  Interventions: Drug: TCMCB07

INTERVENTIONS:
Drug: TCMCB07 — TCMCB07 is will be provided in single-use vials for subcutaneous administration
  Arms: TCMCB07 12.5 mg administered subcutaneously daily for 12 weeks; TCMCB07 25 mg administered subcutaneously daily for 12 weeks; TCMCB07 50 mg administered subcutaneously daily for 12 weeks
Drug: Placebo — Matching placebo
  Arms: Placebo administered subcutaneously daily for 12 weeks

SUMMARY:
This is a randomized, double-blind, placebo-controlled study of B07, administered daily by subcutaneous (SC) injection, in up to 120 patients with newly diagnosed metastatic colorectal cancer. This study will evaluate different doses of B07 on weight, body composition and BMI in patients with sub-optimal BMIs (≤ 29 kg/m^2). Treatment will start at the second cycle of first-line cancer chemotherapy and continue for 12-weeks with the goal of maintaining body weight and muscle mass in patients undergoing chemotherapy relative to control.

ELIGIBILITY:
Inclusion Criteria:

1. Must be at least 18 years of age.
2. An ECOG performance status of ≤ 2.
3. Life expectancy of ≥ 9 months.
4. Able to eat and digest food normally. Patients with colostomies are allowed.
5. Must meet the following:

   1. Newly diagnosed metastatic colorectal adenocarcinoma and about to start first line chemotherapy.
   2. Determined by the Investigator to be ready to receive their second dose of chemotherapy.
6. Starting chemotherapy routines allowed are: FOLFOX, FOLFIRI, or FOLFIRINOX with or without bevacizumab, or other monoclonals or other FDA approved agents to be dosed every 2 weeks. The primary cancer therapy (dose, schedule, or drugs) may be changed as medically indicated.
7. Must have a BMI ≤ 29 kg/m^2.
8. Must be able and willing to safely self-inject daily or be injected by a caregiver.
9. Must have measurable disease by RECIST 1.1 criteria.
10. Must have adequate end organ function as defined by:

    1. ANC ≥ 1.5 × 10^9/L
    2. Platelets ≥ 100 × 10^9/L, or adequate as determined by the medical judgement of the investigator
    3. Hemoglobin ≥ 9 g/dL, or adequate as determined by the medical judgement of the investigator
    4. AST and ALT ≤ 3 × ULN; if liver metastases, then ≤ 5 ×ULN
    5. Bilirubin ≤ 1.5 × ULN or ≤ 3 × ULN in the presence of documented Gilbert's Syndrome
    6. Albumin between 3.4 and 5.4 gm/dL or within institutional normal limits, or not considered clinically significant by the investigator
    7. Creatinine clearance ≥ 50 mL/min (calculated by Cockcroft and Gault equation
    8. Normal hemoglobin A1c levels based on institutional normal limits, or not considered clinically significant by the investigator
11. NT-Pro-BNP and Troponin (TnI or TnT) are within normal limits or not considered to be clinically significant by the investigator.
12. If a female of childbearing capability, must have a negative pregnancy test within 2 weeks of starting treatment.
13. Fertile men and women must agree to use adequate contraception for the duration of the trial.
14. Willing and able to sign informed consent.

Exclusion Criteria

1. Patients receiving second line or later systemic treatment for stage IV disease.
2. Patients with swallowing abnormalities, malabsorption syndromes, short or inflammatory bowel syndromes, or other conditions that in the Investigator's opinion could impair food consumption or metabolism.
3. History of weight loss surgery including gastric stapling, or bypass surgery.
4. Unintentional weight loss ≥ 10% of usual body weight in 4 months prior to Screening or other weight loss considered significant by the Investigator.
5. Currently using any new agent designed to increase appetite or otherwise affect weight (increase or decrease).

   1. THC containing agents (e.g., dronabinol, cannabis). Chronic (> 6 months) use is allowed for THC.
   2. Other weight promoting agents including androgenic compounds (e.g., testosterone, oxandrolone), dopamine antagonists, or megestrol acetate within the past 6 months is excluded.
   3. Newly prescribed glucocorticoids for less than four weeks at the time of Screening and whose weight is not yet stable are excluded. Stable (dose unchanged for 4 weeks or more) and low dose (<4 mg) corticosteroids are permissible, as are inhaled corticosteroids.
6. Chronic and ongoing use of corticosteroids at a dose of ≥5 mg of prednisone or equivalent per day.
7. History of bulimia or anorexia.
8. Pregnancy, lactation, or plans to become pregnant.
9. History of another malignancy except basal cell carcinoma of the skin, carcinoma in situ of the cervix, or other noninvasive or indolent malignancy that has previously undergone potentially curative therapy.
10. Concurrent participation in any other clinical trial.
11. Patients with known brain or CNS metastases.
12. Impaired cardiac function or significant cardiac issues including, but not limited to, any of the following:

    1. Greater than class II NYHA congestive heart failure
    2. Congenital long QT syndrome
    3. QTc > 470 msec (as calculated by institution standards) confirmed by two ECGs ≥ 1-minute apart (interval corrected using [Bazett's formula [QTcB])
    4. Unstable angina pectoris
    5. Acute myocardial infarction ≤ 6 months prior to study entry
13. Known hypersensitivity to B07 or its formulation.
14. Known diagnosis of HIV infection (HIV testing is not mandatory). Patients with a history of HIV regardless of viral load are excluded.
15. Active infection with Hepatitis B, Hepatitis C, or active systemic viral disease or active severe infection.
16. Unwilling or unable to comply with the protocol.
17. Any condition that, in the Investigator's opinion, would impair the patients' ability to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in body weight | At 12 weeks of treatment
Incidence and severity of adverse events (AEs) | From enrollment to the end of the 12 week dosing period
Incidence of abnormalities in laboratory evaluations | From enrollment to the end of the 12 week dosing period
Incidence of abnormalities in vital signs | From enrollment to the end of the 12 week dosing period

SECONDARY OUTCOMES:
Change from baseline in total score of Functional Assessment of Anorexia/Cachexia Therapy-anorexia-related symptoms scale (FAACT-5IASS) | At 12 weeks of treatment
  FAACT-5IASS scores items using a 5-point scale (0-4).Higher scores are associated with a higher health-related quality of life.
Change from baseline in the anorexia and cachexia subscore of the Functional Assessment of Anorexia-Cachexia Therapy (FAACT-ACS) questionnaire | At 12 weeks of treatment
  FAACT-ACS score sums 12 items; both use a 5-point scale (0-4).Higher scores are associated with a higher health-related quality of life.
Change from baseline in BMI | At 12 weeks of treatment
  Weight and height will be combined to report BMI in kg/m^2
Change from baseline in body weight | At 8 weeks of treatment
Change from baseline in BMI | At 8 weeks of treatment
  Weight and height will be combined to report BMI in kg/m^2
Change from baseline in body weight | At 4 weeks of treatment
Change from baseline in BMI | At 4 weeks of treatment
  Weight and height will be combined to report BMI in kg/m^2
Change from baseline in the FAACT questionnaire comprising the general quality of life FAACT-G and FAACT-ACS anorexia and cachexia related subscale | At 12 weeks of treatment
  FAACTG and FAACT ACS score score items using a 5-point scale (0-4).Higher scores are associated with a higher health-related quality of life.
Change from baseline in total score and subscores of European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | At 12 weeks of treatment
  Scoring ranges from 0 to 100 with 0 being the worst possible score and 100 being the best.

OTHER OUTCOMES:
Blood levels of B07 | From enrollment to the end of the 12 week treatment period
  A single blood sample will be taken prior to dose during clinic visits to measure the Cmin blood level of B07
Immunogenicity profile of B07 | From enrollment to the end of the 12 week treatment period
Change from baseline in lean mass | From enrollment to the end of the 12 week treatment period
  Determined by medical imaging
Change from baseline in fat mass | From enrollment to the end of the 12 week treatment period
  Determined by medical imaging
Change from baseline in tumor burden | At 12 weeks of treatment
  To determine the response rate by RECIST 1.1 criteria
Effect of B07 on chemotherapy relative dose intensity | From enrollment to the end of 12 week treatment period
  Comparison of actual dose intensity ratio versus expected chemotherapy dose intensity ratio between B07 and placebo groups

CONTACTS AND LOCATIONS:
Locations (16):
- United States (15):
  - Investigative Site, Tucson, Arizona
  - Investigative Site, Los Angeles, California
  - Investigative Site, Hialeah, Florida
  - Investigative Site, Margate, Florida
  - Investigative Site, Miami Beach, Florida
  - Investigative Site, Tamarac, Florida
  - Investigative Site, Atlanta, Georgia
  - Investigative Site, Wichita, Kansas
  - Investigative Site, Detroit, Michigan
  - Investigative Site, Lincoln, Nebraska
  - Investigative Site, Omaha, Nebraska
  - Investigative Site, Durham, North Carolina
  - Investigative Site, Oklahoma City, Oklahoma
  - Investigative Site, Kingwood, Texas
  - Investigative Site, Laredo, Texas
- Investigative Site, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No